CLINICAL TRIAL: NCT05534620
Title: An Open-label, Non-randomized, Prospective Trial to Evaluate the Effect of Renal Function Impairment and Race/Ethnicity on Treosulfan Pharmacokinetics in Patients With AML or MDS Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Effect of Moderate Renal Impairment and Race/Ethnicity on Treosulfan Pharmacokinetics
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: medac GmbH (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MC-FludT.19/PK
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukaemia (AML); Myelodysplastic Syndrome (MDS); Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Keywords: Pharmacokinetic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — treosulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treosulfan and Fludarabine (Experimental): Participants will receive treosulfan 10 gram per square meter (g/m^2), intravenous (IV) infusion, given over 2 hours once daily on three consecutive days (day -4 to day -2), followed by fludarabine, 30 milligram per square meter (mg/m^2) IV infusion once daily on 5 consecutive days (days -6 to -2), preceding allogeneic haematopoietic stem cell transplantation (alloHSCT) on Day 0.
  Interventions: Drug: Treosulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Treosulfan — IV infusion
Drug: Fludarabine — IV infusion

SUMMARY:
This study aim is to assess, if treosulfan pharmacokinetics are influenced by declined renal function and by race/ethnicity of patients. The study also aims to determine an appropriate safe dose of treosulfan, when patient's renal function is impaired. The participants of this study are undergoing allogenic hematopoietic stem cell transplantation for treatment of acute myeloid leukemia or myelodysplastic syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with AML or MDS who qualify for treosulfan-based conditioning treatment, indicated for alloHSCT.
2. Have available matched-related, matched-unrelated, haploidentical, or a mismatched unrelated donor. Match is defined as at least 9/10 allele matches in human leucocyte antigen (HLA)-A, -B, -C, -DRB1 and DQB1 or 7/8 allele matches in (HLA)-A, -B, -C and -DRB1. Haploidentical is defined as any family member with 2, 3 or 4 (out of 8) HLA-loci mismatch; at the same time, the donor and recipient must be HLA identical for at least one antigen at the following genetic loci: (HLA)-A, -B, -C, and -DRB1. High resolution deoxyribonucleic acid (DNA) typing must be used.
3. Are adults of either sex, age 18-80 years (inclusive).
4. Have a Karnofsky Index of greater than or equal to (>=) 60 percent (%).
5. Have a creatinine clearance (CLcre) >=30 milliliters per minute (mL/min) (Cockcroft Gault: normal renal function: CLcre >=90 mL/min, mild renal impairment: CLcre 60-89 mL/min, moderate renal impairment: CLcre 30-59 mL/min).
6. Are willing to consent to using a highly effective method of birth control, such as condoms, implants, injectables, combined oral contraceptives, intrauterine devices, sexual abstinence or vasectomised partner while on treatment and for at least 6 months thereafter, if females of childbearing potential (defined according to the Clinical Trials Facilitation and Coordination Group guidelines as a fertile woman, following menarche and until becoming postmenopausal unless permanently sterile) and males capable of reproduction.
7. Have a negative pregnancy test, if females of childbearing potential.
8. Have provided a written informed consent.

Exclusion Criteria:

1. Participants considered not eligible for alloHSCT, for instance due to severe concomitant illness, within 3 weeks before the scheduled Baseline Visit:

   * Have severe renal impairment, example, are on dialysis, have renal transplantation history, or calculated CLcre of less than (<) 30 mL/min.
   * Have severe pulmonary impairment, single-breath diffusion capacity of the lung for carbon monoxide (DLCO) (haemoglobin adjusted) or forced expiratory volume (FEV1) of <50%, or severe dyspnoea at rest or requiring oxygen supplementation.
   * Have moderate or severe hepatic impairment (Child-Pugh B or C classification, respectively) and with documented medical history of chronic liver disease..
2. Have a known coronary artery disease, history of myocardial infarction, cardiac dysfunction, including cardiomyopathies, heart failure (New York Heart Association Class II and above), and cardiac arrhythmias (including paroxysmal and permanent atrial fibrillation), interventricular conduction delay and / or bundle branch block (QRS duration >120 milliseconds [ms]).
3. Have Fredericia-corrected QTc (QTcF) interval >450 ms in men and >470 ms in women.
4. Have active malignant involvement of the central nervous system.
5. Are human immunodeficiency virus (HIV) positive or have an active non controlled infectious disease under treatment including fungal infection, active viral liver infection, or known severe acute respiratory syndrome coronavirus 2 (SARS CoV 2) viral infection at the time of enrolment.
6. Have previously had more than one alloHSCT.
7. Have pleural effusion or ascites of >1.0 liters (L).
8. Are pregnant or breast-feeding.
9. Have uncontrolled or severe intercurrent medical condition.
10. Have known hypersensitivity to treosulfan, fludarabine, and / or related ingredients, Fanconi anaemia and other disorders resulting from DNA repair disorders.
11. Are participating in another experimental drug trial (except those for coronavirus disease [COVID 19] vaccines) within 4 weeks prior to the Day 7 Baseline Visit. This exception serves to comply with subject's interests as this population is at a high risk of COVID 19 complications, if the disease occurs. COVID 19 vaccination details (including vaccine name, batch and manufacturer, dose, date of administration, and whether the right or left arm was injected) should be captured as a concomitant medication to enable better assessment of the overall effect of COVID 19 vaccination on oncology trial results.
12. Exhibit non cooperative behaviour or non compliance.
13. Have psychiatric diseases or conditions that might compromise the ability to give informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Area Under the Concentration-time Curve From Time of Administration to the Last Measurable Concentration (AUClast) for Treosulfan | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Area Under the Concentration-time Curve From Time of Administration to Time of Infinity (AUCinf) for Treosulfan | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Area Under the Concentration-time Curve From Time of Administration to the Last Measurable Concentration (AUClast) for Treosulfan Metabolite (Treosulfan Monoepoxide) | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Area Under the Plasma Concentration-time Curve From Time of Administration to Time of Infinity (AUCinf) for Treosulfan Metabolite (Treosulfan Monoepoxide) | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Time to Maximum Observed Plasma Concentration (Tmax) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Time to Last Quantifiable Concentration (Tlast) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Renal Clearance (CL) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Volume of Distribution (Vd) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Terminal Elimination Half-life (t1/2) for Treosulfan and its Metabolite Treosulfan Monoepoxide | Day -4 and Day -2: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Area Under the Concentration-time Curve From Time of Administration to 24 hours (AUC0-24) for Treosulfan and its Metabolite Treosulfan Monoepoxide | At Day -4: Pre-dose, at end of infusion and at 2.5, 3, 4, 6, 8, 12, and 24 hours post-dose
Number of Participants With Engraftment With Treosulfan-based Therapy in Moderate Renal Impairment | Day 0 to Day 28
  Time to engraftment is defined as the time between Day 0 and neutrophil/leukocyte/platelet engraftment. Engraftment includes Neutrophil engraftment, Leukocyte engraftment and Platelet engraftment. Neutrophil engraftment is defined the first of 3 consecutive days with an absolute neutrophil count (ANC) greater than (>) 0.5*10^9 per liter (/L) in peripheral blood (PB) in the first of 3 consecutive days ;Leukocyte engraftment is defined as the first of 3 consecutive days with a total leukocyte count of more than 1*10^9/L in PB. Platelet engraftment is defined as the first of 3 consecutive days with a platelet count of at least 20*10^9/L or of at least 50*10^9/L in PB in the absence of platelet transfusion. Consecutive days is defined as 3 consecutive blood samples, if these are taken on different days.
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Day -7 to Day 28
  A TEAE is defined as any Adverse Event (AE) that has an onset on or after the first dose of investigation medicinal product (IMP) or any pre existing condition that has worsened on or after the first dose of IMP. An SAE or serious adverse reaction (SAR) is any untoward medical occurrence that at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is another medically important event.

CONTACTS AND LOCATIONS:
Overall Officials: Ute Eckenbach, Study Director — SyntheractHCR
Locations (4):
- United States (4):
  - University of Illinois, Chicago, Illinois
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University, Columbus, Ohio
  - VCU Massey Cancer Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No